CLINICAL TRIAL: NCT03477448
Title: The Efficacy of Intra-lesional Bleomycin Versus Intra-lesional Purified Protein Derivative in Treatment of Palmoplantar Warts
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariem Refaat, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Bleomycin Vs PPD
Record Dates: First submitted 2018-03-12; First posted 2018-03-26 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Warts
MeSH Terms: conditions — Warts | interventions — Bleomycin; Tuberculin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PPD group (Active Comparator): This group will include 20 patients who will be treated with IL injection of PPD at a dose of 10 IU (0.1 ml) supplied an insulin syringe in the largest wart.
  Injections will be repeated for all patients into the same lesion (largest wart) every 2 weeks for three treatment sessions
  Interventions: Drug: Purified Protein Derivative
- Bleomycin group (Active Comparator): This group will include 20 patients who will be treated with IL injection of bleomycin.
  Injections will be repeated for all patients into the same lesion (largest wart) every 2 weeks for three treatment sessions, if needed.
  Interventions: Drug: Bleomycin

INTERVENTIONS:
Drug: Bleomycin — an antibiotic derived from Streptomyces verticillus, has an antitumor, antibacterial, and antiviral activity that may be related to its ability to bind with DNA, causing bleomycin strand scission and elimination of pyrimidine and purine bases. The bleomycin hydrolase enzyme, which is known to inactivate bleomycin, is normally found in all body tissues but is present in very small amounts in skin .
  * Intra-lesional bleomycin injection (IBI) has been used for the treatment of warts.
  Arms: Bleomycin group
Drug: Purified Protein Derivative — is an extract of Mycobacterium tuberculosis and is used for testing exposure to tuberculin protein, either from a previous vaccination or from the environment. It contains live, attenuated Mycobacterium bovis.
  * Using this protein derivative for immunotherapy of warts is important for two major aspects. First, because the obligatory immunization program in many developing countries - with high prevalence of wart in many of them - includes BCG vaccination. PPD has a high prevalence of immunity in the general population. Second, although immunotherapy is generally an inexpensive method of treatment in wart patients, PPD, among conventionally used antigens, is the cheapest
  Arms: PPD group

SUMMARY:
* Warts are common viral infections on the skin and are prevalent worldwide. Warts are caused by the human Papilloma virus (HPV), which has more than 100 strains; some of them are known to be premalignant. Although warts can appear at any age, they are more common in children and adolescents. The prognosis of warts cannot be predicted. In some patients they may spontaneously disappear, whereas others show persistence and progression with spreading to other body sites, leading to physical and emotional distress to the patients.
* Factors that increase the risk include use of public showers, working with meat, eczema, and a low immune system . The virus is believed to enter the body through skin that has been damaged slightly . A number of types exist including: common warts, plantar warts, filiform warts, and genital warts . Genital warts are often sexually transmitted.

DETAILED DESCRIPTION:
* Selection of the most appropriate means of treatment is usually difficult because of the availability of various therapeutic lines and also due to the variability in the immune status of the patients for treatment of warts.
* There are on two main therapeutic options: the first is the conventional destructive and aggressive method, which includes treatment with chemical cautery, cryo- therapy, electro cauterization, surgical excision, and laser ablation . This method depends on destruction of the area of epidermis infected with the virus. The recurrence rates after these therapy modalities maybe high. The second is the immunotherapy, which is based on the activation of the immune system to deal with the virus and suppress its activity. Such therapy may be applied either topically or through intra- lesional injection or through systemic administration .
* Intra-lesional immunotherapy utilizes the ability of the immune system to mount a delayed-type hypersensitivity response to various antigens and also the wart tissue. This therapy has been found to be associated with the production of Th1 cytokines that activate cytotoxic and natural killer cells to eradicate HPV infection. This clears not only the local warts but also distant warts, unlike traditional wart therapies .
* Many authors have used different immunotherapeutic agents for intralesional injection. These include Candida antigen, mumps antigen, trichophytin skin test antigen, BCG vaccine, measles, mumps, and rubella (MMR) vaccine, Mycobacterium w (Mw) vaccine, and IFN-α and IFN-γ injectio).
* Bleomycin, an antibiotic derived from Streptomyces verticillus, has an antitumor, antibacterial, and antiviral activity that may be related to its ability to bind with DNA, causing bleomycin strand scission and elimination of pyrimidine and purine bases. The bleomycin hydrolase enzyme, which is known to inactivate bleomycin, is normally found in all body tissues but is present in very small amounts in skin.
* Intra-lesional bleomycin injection (IBI) has been used for the treatment of warts. Numerous reports have been published on the use of intra-lesional bleomycin for the treatment of recalcitrant warts with cure rates ranging from 14 to 99%. It was found to be very effective in treating warts particularly in periungual and palmoplantar areas .
* No systemic side effects have been observed. However, local signs such as necrosis, pain, scaring, pigment change, Raynaud's phenomenon, and nail dystrophy may occur in some cases.
* Purified protein derivative (PPD) is an extract of Mycobacterium tuberculosis and is used for testing exposure to tuberculin protein, either from a previous vaccination or from the environment. It contains live, attenuated Mycobacterium bovis.
* Using this protein derivative for immunotherapy of warts is important for two major aspects. First, because the obligatory immunization program in many developing countries - with high prevalence of wart in many of them - includes BCG vaccination. PPD has a high prevalence of immunity in the general population. Second, although immunotherapy is generally an inexpensive method of treatment in wart patients, PPD, among conventionally used antigens, is the cheapest.
* IL purified protein derivative (PPD) injection is an acceptable and safe modality in the treatment of warts with complete response in 75% of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with positive tuberculin test or with past history of PPD vaccination will include.
* Patient with normal CBC , liver function and renal function

Exclusion Criteria:

* Patients with immunosuppression, pregnancy, or lactation, with negative tuberculin test or with past history of tuberculosis, peripheral vascular disease, any abnormality in liver or renal function and those who received any wart treatment 1 month before the start of the study will exclude.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
The cure rate of patients | One year
  the clinical disappearance of the warts

REFERENCES:
- [Background] Lynch MD, Cliffe J, Morris-Jones R. Management of cutaneous viral warts. BMJ. 2014 May 27;348:g3339. doi: 10.1136/bmj.g3339. No abstract available. PMID 24865780
- [Background] Yamamoto T. Bleomycin and the skin. Br J Dermatol. 2006 Nov;155(5):869-75. doi: 10.1111/j.1365-2133.2006.07474.x. PMID 17034512